CLINICAL TRIAL: NCT01610544
Title: A Pilot Study of 18F FLT PET/CT in Evaluating Early Response to Anti-Proliferative Therapies in Non Small Cell Lung Cancer and Thymic Tumors
Brief Title: 18F FLT Imaging Studies of Treatment Response for Lung Cancer and Thymoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 120130; 12-C-0130
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-12-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Thymus Neoplasms
Keywords: Thymoma; Insulin Growth Factor; Cell Proliferation; Non Small Cell Lung Cancer; PET/CT Imaging Sessions
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Thymus Neoplasms; Thymoma; Hyperplasia | interventions — alovudine

INTERVENTIONS:
Drug: 3'-deoxy-3'-18F fluorothymidine (FLT)
Other: PET/CT scan

SUMMARY:
Background:

- Imaging studies like positron emission tomography (PET) and computed tomography (CT) scans are used to detect tumor responses to cancer treatment. However, it may be difficult to detect early response to lung cancer or thymoma treatment with standard PET/CT scans. These scans cannot easily show a difference between remaining cancer cells and inflammation. Researchers want to try a new PET/CT scan tracer that may be able to show the difference between these cells. 18F-Fluorothymidine (18F-FLT) is better at showing which cells are still actively dividing. PET/CT scans with 18F-FLT may help show if tumor cells are responding to early stages of treatment.

Objectives:

- To see if 18F-FLT is a safe and effective imaging study tracer to show early cancer response to treatment.

Eligibility:

- Individuals at least 18 years of age who are being treated for lung cancer or thymoma.

Design:

* Participants will be screened with a physical exam and medical history. Blood, urine, and tumor tissue samples will be collected.
* Participants will have two PET/CT scans on separate days before starting chemotherapy. One scan will be with a standard radiotracer. The other will be with the 18F-FLT tracer.
* About 2 weeks after starting chemotherapy, participants will repeat the two PET/CT scans on separate days. Additional blood samples will be collected at this time.

DETAILED DESCRIPTION:
Background:

* (18)F FLT, a thymidine analog, has uptake in tumors that correlates with proliferative rates and may be an early predictor of tumor response.
* Due to uptake in inflammatory tissues, routinely used (18)F FDG PET/CT is often unable to distinguish therapeutic response from reactive change early in therapy.
* Molecularly targeted therapies relating to the MEK kinase pathway in non small cell lung cancer (NSCLC) and the IGF pathway (anti-IGF-1R monoclonal antibodies) in thymoma, affect tumor proliferation.
* We intend to explore the potential utility of (18)F FLT PET/CT imaging as an early marker of therapeutic response in molecularly targeted therapies relating to the MEK kinase pathway in NSCLC and the IGF pathway in thymic tumors.

Objectives:

-To explore the relationship between change in (18)F FLT tumor uptake (pre-treatment and soon after initiation of treatment (2 weeks)) and progression free survival in NSCLC patients treated with AZD6244 and in thymoma patients with IMC-A12, Cixutumumab

Eligibility:

* Subjects with pathology proven lung cancer or thymoma enrolled in an NCI therapy protocol.
* Participant must be 18 years or older and have ECOG Performance of less than or equal to 2.
* Patients must have measurable disease by RECIST criteria.
* Patients must have the ability to provide informed consent. All subjects must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

Design:

-This is a pilot study which will incorporate (18)F FLT and (18)F FDG PET/CT imaging sessions prior to therapy with AZD6244, Selumetinib, in NSCLC and IMC-A12, Cixutumumab, in thymoma, and 2 weeks (+/- 4 days) following therapy initiation. The imaging parameters will be evaluated with respect to clinical response (as determined under the referring protocol). We expect to enroll 24 evaluable patients in this single center study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects with pathology proven lung cancer or thymic malignancy already enrolled in an NCI treatment protocol usingAZD6244 in NSCLC and IMC-A12, in thymoma.
* Participant must be 18 years or older
* ECOG Performance score of 0 to 2
* Ability to provide informed consent. All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of this study before any protocol related studies are performed.
* Participants must NOT be pregnant or intend to become pregnant within 1 week of the last injection of (18)F FLT

EXCLUSION CRITERIA:

* Known allergy to fluorothymidine
* Participants for whom enrollment would significantly delay (> 2 weeks) the scheduled standard of care therapy
* Participants with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results are excluded
* Participants with severe claustrophobia not relieved by oral anxiolytic medication or patients weighing >136 kg (weight limit for scanner table)
* Other medical conditions deemed by the PI or associates to make the patient ineligible for protocol procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05-10; Primary Completion 2012-12-10 (Actual); Study Completion 2012-12-10 (Actual)

PRIMARY OUTCOMES:
To explore the relationship between change in 18F FLT tumor uptake and progression free survival in NSCLC patients treated with AZD6244 and in thymoma patients with IMC-A12, Cixutumumab

SECONDARY OUTCOMES:
To explore the relationship between the absolute pre-treatment 18F FLT uptake and the clinical response to therapy
To determine if the change in 18F FLT uptake is different from the change in 18F FDG PET/CT at the same time points

CONTACTS AND LOCATIONS:
Overall Officials: Maria Liza Lindenberg, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] McKian KP, Haluska P. Cixutumumab. Expert Opin Investig Drugs. 2009 Jul;18(7):1025-33. doi: 10.1517/13543780903055049. PMID 19548856
- [Background] Shields AF, Mankoff DA, Link JM, Graham MM, Eary JF, Kozawa SM, Zheng M, Lewellen B, Lewellen TK, Grierson JR, Krohn KA. Carbon-11-thymidine and FDG to measure therapy response. J Nucl Med. 1998 Oct;39(10):1757-62. PMID 9776283
- [Background] Vesselle H, Grierson J, Muzi M, Pugsley JM, Schmidt RA, Rabinowitz P, Peterson LM, Vallieres E, Wood DE. In vivo validation of 3'deoxy-3'-[(18)F]fluorothymidine ([(18)F]FLT) as a proliferation imaging tracer in humans: correlation of [(18)F]FLT uptake by positron emission tomography with Ki-67 immunohistochemistry and flow cytometry in human lung tumors. Clin Cancer Res. 2002 Nov;8(11):3315-23. PMID 12429617